CLINICAL TRIAL: NCT06674421
Title: Reliability of GYKO Inertial Sensor System in the Assessment of Jumping and Postural Stability Parameters in Adolescent Basketball Players
Brief Title: Reliability of GYCO in Basketball Players
Status: Not yet recruiting | Type: Observational
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Emel Tasvuran, Assoc. Prof., Sakarya University
Other Study IDs: 49/12
Record Dates: First submitted 2024-11-03; First posted 2024-11-05 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Healthy
Keywords: athletes; validity and reliability; jump; postural stability

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Basketball players: Participants will be adolescent athletes attending the basketball course at Alaağaç Sports Club. Being between the ages of 10-19 years and being playing basketball.
  Interventions: Other: Reliability Analyses

INTERVENTIONS:
Other: Reliability Analyses — For the reliability analysis test-retest method will use. There will be a one-week break between the first test and the retest.

SUMMARY:
The aim of this study was to evaluate the reliability of the GYKO, which enables the assessment of jump and postural stability parameters of athletes, in adolescent basketball players.

DETAILED DESCRIPTION:
GYKO is a device used to evaluate joint function, muscle strength, jumping and postural stability parameters during rehabilitation of a specific region of the musculoskeletal system. The aim of this study was to evaluate the reliability of the GYKO, which enables the assessment of jump and postural stability parameters of athletes, in adolescent basketball players.

The research will be conducted at Sakarya University of Applied Sciences Physiotherapy and Rehabilitation Application and Research Centre. The participants will consist of adolescent athletes attending the basketball course at Alaağaç Sports Club.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 10-19 years old
* Being playing basketball.

Exclusion Criteria:

* Having musculoskeletal system, rheumatological, cardiovascular etc. diseases

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants will be adolescent athletes attending the basketball course at Alaağaç Sports Club.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2024-12-02 (Estimated); Primary Completion 2025-03-03 (Estimated); Study Completion 2025-06-02 (Estimated)

PRIMARY OUTCOMES:
Counter Movement Jump | The evaluation will be conducted at the baseline and 1 week after the first evaluation.
  Counter movement jump height will be assessed by GYKO sensor. The jump height will be saved.

CONTACTS AND LOCATIONS:
Overall Officials: EMEL TAŞVURAN HORATA, Assoc. Prof., Principal Investigator — Sakarya University of Applied Sciences; Oğuzhan Bahadır Demir, PhD, Study Chair — Sakarya University of Applied Sciences; Birgül DINGIRDAN GÜLTEKİNLER, MSc, Study Chair — Sakarya University of Applied Sciences

IPD SHARING:
Plan to Share IPD: No